CLINICAL TRIAL: NCT04244344
Title: A Pilot Fall Prevention Program Using "STRATIFY" at Triage of Emergency Department in Hong Kong
Acronym: Prevent Fall
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, LAU, Wai Yuen, Regestered Nurse, Prince of Wales Hospital, Shatin, Hong Kong
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Prevent Fall in AED
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Intervention for Fall Prevention
Keywords: Intervention; Fall; Fall Prevention

STUDY DESIGN:
Intervention Model Description: The subjects who meet the criteria of high fall risk using "STRATIFY' tool will receive several fall preventions in order to prevent their fall incidence, survey will be conducted to gether their opinion about the interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional (Experimental): all High fall risk subjects who meet the criteria by "STRATIFY" Tool
  Interventions: Other: fall prevention measures

INTERVENTIONS:
Other: fall prevention measures — High fall risk signage, information sheet, High fall risk bracelet, verbal instructions

SUMMARY:
A fall is an event which results in a person coming to rest unwittingly on the floor or ground or other lower level. Those who have fall history have significantly more hospitalizations and clinical visits as well as emergency department visits than those who do not. Loss of confidence in walking, fear of falling, social isolation and depression can also occur in those patients. Fall is a predictor for decreased functional status and risk factor for the whole institution Approximately 30% to 40% of people aged 65 years and older who lived in the community fall each year. Multiple studies related to falls have shown a close relation between sex and age. As a result, Elderlies who are prone to falling consume more health care resources than non-fallers.

STRATIFY proved to be more accurate and more frequently utilized. STRATIFY was originally derived in mixed acute/rehabilitation geriatric wards of UK urban teaching hospital using a 'case control' design and multi-variate regression to identify predictors of falls in hospital inpatients. This resulted in a simple five-point score (each item scoring 1 or 0), with predictive "cut-offs" as 2 or 3 used in the original validation studies which followed. STRATIFY was not designed or validated for continuous modelling of risk but for use in categorical prediction 'high' versus 'low risk'. Sensitivity and specificity were both found to be in excess of 80% in the two UK cohort of the original paper, leading to wide spread adoption of the tool in clinical practice. It is now ten years since the publication of the original STRATIFY paper and a number of prospective studies in several cohort of patients have been published.

Objective and Propose

1. To assess the effectiveness of the fall preventing intervention after targeted group is screened by the tool "STRATIFY" in triage
2. To look at the discrepancy of fall perception of patient/caregiver and the assessment result using "STRATIFY".
3. To compare the fall rate after applying the screening tool "STRATIFY" and with intervention given in their AEDs.

Hypothesis

1. It is hypothesized that the effectiveness score collected from patient and/or caregivers via questionnaires within data collection period shows positive result and these measures are worth to execute in A&E.
2. It is hypothesized that there may not be a big discrepancy of fall perception of caregivers with the result of assessment tool and there is a discrepancy of fall perception of fall perception of patients as they may over-estimate their ability
3. It is hypothesized that the fall rate of intervention group will be lower than that of control group.

Rate of fall incident which is properly documented and reported to AIRS after using fall screening tool "STRATIFY" and intervention given will be the intervention group.

Rate of fall incident of usual practice in a designated period will be the control group.

DETAILED DESCRIPTION:
Methodology:

Design: Prospective two-center observational study Data collection Frequency: Cross-sectional Sampling Design: convenience sampling Sampling Tool: Assessment forms & Questionnaires

Data collection Time:

Subject recruitment started from 1/2020 to 3/2020. Geriatric Attendance were extracted from the Clinical Data Analysis and Reporting System (CDARS) in the period of 1/2019 to 3/2019 and 1/2020 to 3/2020 Numbers of fall cases were extracted from AIRS system. Setting: KWH A&E and PWH A&E (different cluster)

Population and sample size For a 95% confidence interval with width=0.3, the expected sample size is at least 267 subjects needed to be recruited based on the rule of thumb that SD = range/4. In this study, approximately 300 subjects will be recruited (~150 from Kwong Wah Hospital and ~150 from Prince of Wales Hospital) .

Subject recruitment:

Nurse investigators will be assigned to different duty by Duty in-charge in each shift. First of all, the research nurse will screen the case with inclusion and exclusion criteria. After that, investigators will approach to the target group, 10mins will be given to the target group to consider whether to participate in the study or not. Once the target group decided to participate in the research, fall risk of targeted patients will be screened by using "STRATIFY" fall risk assessment tool at triage by investigators. Patient will be screened into 2 groups, either at risk (score≥2) or not at risk (score<2). Nursing intervention includes fall signage, fall bracelet, instruction card will be provided to high risk group (score≥2). Questionnaires will be distributed to the target groups to collect their opinions towards the screening tool and the intervention upon they were discharged or admitted.

Content Validity The content validity of patient/caregiver effectiveness score questionnaire and instruction card will be established by a panel of eight including one geriatric nursing consultant, one emergency nursing consultant, two emergency medicine specialists and four advanced practice nurses from two A&Es. They will review the questionnaire and all suggestions will be incorporated into the final version of the questionnaire. Ten lay persons will be invited to complete the questionnaire to examine the readability to general public.

Selection and Withdrawal of subjects Nurse investigator will be assigned to different duty by Duty in-charge in each shift. First of all, the research nurse will screen the case with inclusion and exclusion criteria. After that, investigators will approach to the target group, 20mins will be given to the target group to consider whether to participate in the study or not. Once the target group decided to participate in the research, fall risk of targeted patients will be screened by using STRATIFY at triage by investigators. Patient will be screened into 2 groups, either at risk (score≥2) or not at risk (score<2).

Nursing interventions Fall signage, fall bracelet, instruction card will be provided to high risk group. Patients of high risk group will be positioned close to the nurse's station. For high risk patients, nurse should ensure that the bed is at the lowest height, the brakes are locked and the patient's belongings are within reach. Questionnaires will be distributed to the target groups to collect their opinions towards the screening tool and the interventions.

Inclusion criteria:

Patient aged 65years old or above Caregiver aged 18years old or above and has cared patient for at least 1month Able to read and listen Cantonese/English Able to consent Triage category 3, 4, 5 Using Hong Kong Identity Card for registration

Exclusion criteria Patient who has done the fall assessment using Morse Fall Scale (i.e. patient in Observation Ward in KWH and patient who admitted to EM Ward in PWH) Caregivers of patient who has done the fall assessment using Morse Fall Scale Unable to consent Unable to read and listen Cantonese/English Triage category 1&2 cases

Primary Outcome:

The effectiveness score of the fall preventing intervention collected from patient and/or caregivers via questionnaires within data collection period (Questionnaire Q2 & Q4).

Secondary Outcome:

The discrepancy of fall perception of patient/caregiver to STRATIFY screening tool (Questionnaire Q1).

Number of fall cases in A&E of PWH and KWH which are properly documented and reported to AIRS.

Method of Data Analysis The effectiveness score collected from patient and/or caregivers via questionnaires within data collection period (Questionnaire Q1-3) will be presented using descriptive method. The confidence intervals, correlation will be calculated.

The discrepancy of fall perception of patient/caregiver to STRATIFY screening tool (Questionnaire Q4) is analyzed by constructing CI which estimates the proportion of subjects who do not know they are high risk but they actually are.

Number of fall cases in A&E of PWH and KWH which are properly documented and reported to AIRS will be analyzed and presented with descriptive method.

Direct Access to Source Data and Documents The principal investigator and other investigators of the research team are responsible for data collection and they will be permitted to access to source data and study record.

Quality Control and Quality Assurance Daily logs will be recorded by the research nurse to monitor the study progress including the number of respondents approached, interviews completed or refused and incomplete interviews. All data entered in the database will be verified and cleaned. After completion of data entry, computer logic checks will be run for consistency of related code. Questionable data will be reviewed against the hard copy of questionnaire. Necessary corrections will be made to the database.

Ethical approval The protocol will be submitted to the Research Ethics Committee (Kowloon Central/Kowloon East and NTEC). The conduct of the study will be complied with the "declaration of Helsinki". Participation in the study is voluntary and withdrawal is allowed at any moment during data collection. An information sheet is provided and a written consent is required from the participant.

Data Handling, Record Keeping, Publication and Disposal All identifiable personal data will be anonymized and will follow the HA policy on handling of patient data privacy. The completed questionnaires and records will be kept in a locked cabinet for 3 years. The computerized research and personal data will be kept by encryption with restricted use to authorized person only. All data are used for research only.

The completed questionnaires will be destroyed by cross-cut shredding and disposed to confidential disposal container. The computerized research and personal data will be destroyed by data erasure software to ensure the data cannot be recovered. The data disposing procedure will be held at the end of 3 years storage period.

Financing and Insurance Not applicable

Publication Policy The dissemination of research findings will be presented in post registered core course.

Supplements Written consent form, questionnaires and patient information sheet.

Indemnity and Insurance N/A

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65years old or above
* Caregiver aged 18years old or above and has cared patient for at least 1month
* Able to read and listen Cantonese/English
* Able to consent
* Triage category 3, 4, 5
* Using Hong Kong Identity Card for registration

Exclusion Criteria:

* Patient who has done the fall assessment using Morse Fall Scale (i.e. patient in Observation Ward in KWH and patient who admitted to EM Ward in PWH)
* Caregivers of patient who has done the fall assessment using Morse Fall Scale
* Unable to consent
* Unable to read and listen Cantonese/English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The effectiveness score of the fall preventing intervention collected from patient and/or caregivers via questionnaires within data collection period | 3 months
  using the survey to collect data

SECONDARY OUTCOMES:
The discrepancy of fall perception of patient/caregiver to STRATIFY screening tool | 3 months
  using the survey to collect data

CONTACTS AND LOCATIONS:
Locations (1):
- AED, Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
all invertigator can access the data collected
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: will be available in 3 months and will be kept for 3 years
Access Criteria: all investigator and departmatal use when needed

REFERENCES:
- [Background] Chu LW, Chiu AY, Chi I. Falls and subsequent health service utilization in community-dwelling Chinese older adults. Arch Gerontol Geriatr. 2008 Mar-Apr;46(2):125-35. doi: 10.1016/j.archger.2007.03.005. Epub 2007 Apr 27. PMID 17467081
- [Background] Luk JKH, Chiu PKC, Chu LW. Factors affecting institutionalization in older Hong Kong Chinese patients after recovery from acute medical illnesses. Arch Gerontol Geriatr. 2009 Sep-Oct;49(2):e110-e114. doi: 10.1016/j.archger.2008.10.007. Epub 2008 Dec 17. PMID 19095312
- [Background] Phelan EA, Mahoney JE, Voit JC, Stevens JA. Assessment and management of fall risk in primary care settings. Med Clin North Am. 2015 Mar;99(2):281-93. doi: 10.1016/j.mcna.2014.11.004. PMID 25700584
- [Background] Oliver D, Papaioannou A, Giangregorio L, Thabane L, Reizgys K, Foster G. A systematic review and meta-analysis of studies using the STRATIFY tool for prediction of falls in hospital patients: how well does it work? Age Ageing. 2008 Nov;37(6):621-7. doi: 10.1093/ageing/afn203. Epub 2008 Oct 1. PMID 18829693